CLINICAL TRIAL: NCT05715658
Title: A Study Evaluating the Pharmacokinetics of Dabigatran Etexilate in Adult Healthy Subjects, Elderly Healthy Subjects, and Elderly Patients With Atrial Fibrillation
Brief Title: Pharmacokinetic Study to Evaluate Dabigatran Etexilate in Elderly Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dongyang Liu (Other)
Responsible Party: Sponsor-Investigator, Dongyang Liu, Vice director of Drug Clinical Center, Peking University Third Hospital
Organization: Peking University Third Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: M2022280
Record Dates: First submitted 2022-07-04; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Nonvalvular Atrial Fibrillation; Health, Subjective
Keywords: dabigatran pharmacokinetics; P-glycoprotein; older adult
MeSH Terms: interventions — Dabigatran

STUDY DESIGN:
Intervention Model Description: Control group: 12 healthy adults (18-30 years old); Test group A: 12 elderly healthy people (≥75 years old); Test group B: 12 elderly patients with atrial fibrillation (≥75 years old).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Evaluating the pharmacokinetics of dabigatran etexilate in elderly healthy subjects (Experimental): Adult healthy subjects and elderly healthy subjects only took one 110mg dabigatran etexilate capsule orally, and elderly patients with atrial fibrillation took dabigatran etexilate according to routine medical care.
  Interventions: Drug: Dabigatran etexilate capsule

INTERVENTIONS:
Drug: Dabigatran etexilate capsule — Adult healthy subjects and elderly healthy subjects only take one 110 mg dabigatran etexilate capsule (low-dose specification in the instruction manual) orally. Elderly patients with atrial fibrillation take dabigatran etexilate according to routine medical treatment.

SUMMARY:
This study intends to collect blood samples of adult healthy subjects, elderly healthy subjects and elderly patients with atrial fibrillation after taking dabigatran etexilate for pharmacokinetics and other studies, aiming to reveal the effect of dabigatran etexilate in Chinese elderly population. Pharmacokinetic profile and biomarker concentration levels; fecal samples were collected for gut microbiota studies to further explore potential mechanisms. The results of the study may provide reference for the precision medicine of dabigatran etexilate and other drugs in the elderly population or the development of new clinical drugs.

DETAILED DESCRIPTION:
This study is a single-center, open-label clinical study, with adult healthy subjects, elderly healthy subjects and elderly patients with atrial fibrillation as the research subjects. Adult healthy subjects and elderly healthy subjects only take one 110 mg dabigatran etexilate capsule (low-dose specification in the instruction manual) orally. Elderly patients with atrial fibrillation take dabigatran etexilate according to routine medical treatment. Blood samples at 0 h(before dosing), 2 h, 6 h, 10 h and 24 h after dosing, and additional stool samples were collected.

ELIGIBILITY:
Inclusion Criteria:

1. With full capacity for civil conduct, the age of adult healthy subjects is ≥18 years old and ≤30 years old; elderly healthy subjects ≥ 75 years old; elderly patients with atrial fibrillation are ≥75 years old.
2. Male weight ≥ 50 kg, female weight ≥ 45 kg; body mass index (BMI) within the range of 19.0~27.0 (including upper and lower limits), body mass index (BMI) = weight (kg) / height 2 (m2).
3. Creatinine clearance rate (CRCL): calculated by Cock Croft-Gault equation, adult healthy subjects should have CRCL≥90mL/min; elderly healthy subjects should have CRCL≥60mL/min; elderly patients with atrial fibrillation should have CRCL≥30mL/min.
4. Elderly patients with atrial fibrillation should have meet the diagnostic criteria for non-valvular atrial fibrillation.
5. Elderly patients with atrial fibrillation are taking Dabigatran etexilate for routine treatment.

Exclusion Criteria:

1. History of fainting of needles and blood.
2. Diseases affecting intestinal P-glycoprotein: severe diarrhea (excretion more than 3 times a day with watery stool characteristics), Crohn's disease, ulcerative colitis, irritable bowel syndrome, diverticulitis, difficult Identify Clostridium infection (recurrent) or Helicobacter pylori infection.
3. Diseases affecting the activity of CYP3A in the liver: acute kidney injury, liver cirrhosis, liver abscess, liver cancer, intrahepatic bile duct stones, etc.
4. Diseases affecting changes in intestinal flora: non-alcoholic fatty liver disease, diabetes, chronic constipation.
5. History of major diseases or newly discovered diseases: prostate cancer, leukemia, liver cancer, breast cancer, colorectal cancer, leukemia and other tumor diseases.
6. Diseases or conditions with significant risk of major bleeding, such as current or recent peptic ulcer, malignant neoplasms with high bleeding risk, recent brain or spinal cord injury, recent brain, spinal cord, or eye surgery, recent intracranial hemorrhage, known or suspected Esophageal varices, arteriovenous malformations, vascular aneurysms, or major intraspinal or intracranial vascular abnormalities.
7. Clinically significant active bleeding.
8. Are using anticoagulant drugs such as unfractionated heparin (UFH), low molecular weight heparin (LMWH) and heparin derivatives (fondaparinux sodium), vitamin K antagonists, rivaroxaban or other direct thrombin Inhibitors (recombinant hirudin, bivalirudin); thrombolytic drugs; or current use of antiplatelet aggregation drugs such as GPIIb/IIIa receptor antagonists, ticlopidine, prasugrel, dextran, sulfinpyrazone, aspirin, etc.
9. Use of drugs that may affect the intestinal flora within 1 week before the trial: Continuous use of antibiotics, Bifidobacterium triple viable bacteria powder, lactobacillus tablets, compound Lactobacillus acidophilus tablets, Bacillus subtilis dual viable bacteria enteric-coated capsules, containing bismuth subsalicylate, etc.
10. Use of drugs that may affect the activity of intestinal P-glycoprotein/CYP3A within 1 week before the trial: ① Potent P-glycoprotein/CYP3A inhibitors: amiodarone, verapamil, diltiazem, quinidine, dronedarone, tacrolimus, cyclosporine, protease inhibitors indinavir, nelfinavir, saquinavir, lopinavir), macrolide antibiotics (erythromycin, clarithromycin, telithromycin), chloramphenicol, azole Antifungal drugs (ketoconazole, itraconazole, Posaconazole, voriconazole, fluconazole, miconazole), nefazodone, cobicistat, cimetidine, ciprofloxacin, Imatinib, St. John's Wort, Ranolazine; ② Potent P-glycoprotein/CYP3A inducers: rifampicin, carbamazepine, phenytoin, phenobarbital, dexamethasone, antiandrogens (enzalutamide, apalutamide).
11. Those who have a history of smoking and drinking in the past, and who do not agree with the prohibition of smoking and drinking during the trial period: smokers (the average daily cigarettes smoked more than 5 cigarettes within one month before the test); alcoholism (the average daily drinking within one month before the test) ≥100mL high-quality liquor (ethanol content ≥40%)).
12. History of gastrointestinal surgery such as gallbladder or appendectomy, bariatric surgery, etc. within the past 6 months.
13. Positive virological test (human immunodeficiency virus antibody (HIV-Ab), syphilis serological test, hepatitis B virus surface antigen (HBsAg) or hepatitis C virus antibody (HCV-Ab)) within 3 months before screening.
14. Those who have participated in clinical trials of any drug or medical device within 1 month before screening (in the case of drug clinical trials, those who participated in the previous clinical trial before screening have more than 5 half-lives).
15. Subjects who are considered by the investigator to have any factors that are not suitable for participating in this trial.

    Adult healthy subjects, with the following additional exclusion criteria:
16. Pregnant and lactating women.
17. Suffering from atrial fibrillation, hypertension, heart failure, coronary heart disease, heart valve disease and other diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Concentration in plasma of dabigatran on the first day before administration | on the first 1 day before administration
  Plasma concentration of dabigatran will be measured by LC-MS/MS or HPLC
Concentration in plasma of dabigatran on the 2, 6, 10, and 24 hours after administration | on the 2, 6, 10, and 24 hours after administration
  Plasma concentration of dabigatran will be measured by LC-MS/MS or HPLC
Species of intestinal flora | on the first 1 day before administration
  Bacterial composition will be measured by 16s or Metagenome

SECONDARY OUTCOMES:
Gene polymorphsim | on the first 1 day before administration
  Gene polymorphisms of CES1, CES2, P-glycolprotein will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Dongyang Liu, Principal Investigator — Drug Clinical Trial Center
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hines LE, Murphy JE. Potentially harmful drug-drug interactions in the elderly: a review. Am J Geriatr Pharmacother. 2011 Dec;9(6):364-77. doi: 10.1016/j.amjopharm.2011.10.004. Epub 2011 Nov 11. PMID 22078863
- [Result] Zorab PA. Proceedings: Prognosis for life in childhood scoliosis. Arch Dis Child. 1973 Oct;48(10):824-5. doi: 10.1136/adc.48.10.824-c. No abstract available. PMID 4749689
- [Result] Elmeliegy M, Vourvahis M, Guo C, Wang DD. Effect of P-glycoprotein (P-gp) Inducers on Exposure of P-gp Substrates: Review of Clinical Drug-Drug Interaction Studies. Clin Pharmacokinet. 2020 Jun;59(6):699-714. doi: 10.1007/s40262-020-00867-1. PMID 32052379